CLINICAL TRIAL: NCT05671926
Title: Different Algorithm Models to Predict Postoperative Pneumonia in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: PPC2021012
Record Dates: First submitted 2023-01-02; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pulmonary Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training set: The whole cohort is randomly assigned to a training cohort and validation cohort.
- validation set: The whole cohort is randomly assigned to a training cohort and validation cohort.

SUMMARY:
The researchers aim to compare different algorithms to predict postoperative pneumonia in elderly patients and to assess the risk of pneumonia in elderly patients.

DETAILED DESCRIPTION:
Postoperative pneumonia is a common complication that increases the mortality and length of older patients. In order to better assess the risk of postoperative pneumonia in elderly patients, we plan to use database information and different algorithms, such as logistic regression, random forest, and other algorithms respectively to build models and evaluate the effects of the models.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. receiving invasive ventilation during general anesthesia for surgery

Exclusion Criteria:

1. preoperative mechanical ventilation
2. procedures related to a previous surgical complication
3. a second operation after surgery
4. organ transplantation
5. discharged within 24 hours after surgery
6. cardiac and thoracic surgery

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: older patients received general anesthesia in Wuhan Union Hospital from January 1, 2014 to December 31, 2019.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | within one week after surgery

SECONDARY OUTCOMES:
Postoperative pulmonary complications | 30 days after surgery